CLINICAL TRIAL: NCT02654665
Title: Comparing Effects of Liraglutide and Bariatric Surgery on Weight Loss, Liver Function, Body Composition, Insulin Resistance, Endothelial Function and Biomarkers of Non-alcoholic Steatohepatitis (NASH) in Obese Asian Adults
Acronym: CGH-LiNASH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Joan Khoo Joo Ching, Chief & Senior Consultant, Changi General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGH-LiNASH
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Weight Loss; Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liraglutide (Experimental): Liraglutide will be administered once daily by subcutaneous injection at a starting dose of 0.6 mg, increasing at 0.6 mg/week increments to a maximum of 3.0 mg over the next 6 weeks, as tolerated.
  Interventions: Behavioral: Lifestyle modification
- Bariatric Surgery (Active Comparator): Subjects will have outcomes measured within 28 days before surgery. Post-operative management and frequency of follow-up visits will be decided by the bariatric surgeon. Study visits for biochemical and endothelial function testing; MRI and liver biopsy and / or fibroscan will follow the same schedule as that of the lifestyle and liraglutide arms. Target weight loss for the first 26 weeks post-surgery is at least 30% of excess body weight.
  Interventions: Drug: Liraglutide
- Diet modification and exercise (Active Comparator): Exercise will be used to induce and maintain weight loss in a 26-week Weight Management Program. Each subject will follow an aerobic exercise prescription of moderate intensity (60-75% maximum heart rate) to expend 2000-3000 kcal/week, lasting 30-60 minutes each session (over 5-7 sessions). Subjects will be instructed by sports trainers, compliance reviewed and adjusted if necessary to maintain the targeted total energy expenditure to produce weight loss of at least 7% over 26 weeks.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Behavioral: Lifestyle modification — Diet and exercise designed for 5-7% weight loss over 6 months
  Arms: Liraglutide
Drug: Liraglutide — GLP-1 agonist
  Other Names: Victoza
  Arms: Bariatric Surgery; Diet modification and exercise

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is defined by presence of hepatic steatosis (fat accumulation in liver cells), either by imaging or by biopsy and absence of causes for secondary hepatic fat accumulation such as significant alcohol consumption, medications, or hereditary disorders. In the majority of patients, NAFLD is associated with risk factors for cardiovascular disease such as obesity, diabetes mellitus, and high cholesterol, and may lead to irreversible liver damage. Non-alcoholic steatohepatitis (NASH) is a more severe form of NAFLD and is present in up to 30% of obese adults. NASH is defined by hepatic steatosis and inflammation with hepatocyte injury with or without fibrosis (hardening of the liver).

The prevalence, morbidity and mortality of NAFLD is increasing, particularly in the Asia-Pacific region where there will be an estimated 300 million obese people by 2030. Weight loss is the first-line treatment for NAFLD in obese individuals, but the utility of lifestyle modification with diet and exercise is limited by difficulties in sustaining compliance and by eventual weight regain. Bariatric (weight loss) surgery produces the greatest amount of weight loss but is limited by cost, patient acceptance, and complications. The efficacy of drugs for NASH, such as vitamin E and medication to lower cholesterol and glucose, remains unclear. Liraglutide, a glucagon-like peptide (GLP-1) analogue, is an injectable medication which has been shown to induce weight loss and lower glucose in obese adults. There is little information on the effects of GLP-1 analogues on NASH, particularly in comparison to other modalities of weight loss such as surgery. This study aims to compare the efficacy and safety of lifestyle modification, liraglutide and surgery, for weight loss in conjunction with reducing severity of NASH, and for insulin resistance, high cholesterol and other cardiovascular risk factors.

DETAILED DESCRIPTION:
The morbidity and mortality from non-alcoholic fatty liver disease (NAFLD), the most common liver disease worldwide, are rapidly increasing as a result of the global explosion in obesity, particularly in the Asia-Pacific region where there will be an estimated 300 million obese people by 20302. Non-alcoholic steatohepatitis (NASH), a subset of NAFLD, which is present in up to 30% of obese adults, leads to irreversible liver cirrhosis, and is associated with type 2 diabetes, cardiovascular disease and increased morbidity and mortality. Weight loss has established efficacy on NASH-associated cardiometabolic abnormalities and disease activity and severity. Diet and exercise produce a modest effect on NASH which is limited by weight regain, even with intensive lifestyle modification. Bariatric surgery produces the greatest amount of weight loss, but is less acceptable to many patients than lifestyle modification or medical therapy, and is limited by cost and complications, particularly post-surgical malabsorption and potential psychological complications. The efficacy of previously-studied medications on NASH, such as statins, insulin sensitizers and ursodeoxycholic acid, remains unclear.

This study therefore aims to compare the efficacy and safety of a medication which induces weight loss and reduces insulin resistance, with that of lifestyle modification (diet and exercise), and bariatric surgery, for improvement in NASH severity, insulin resistance and other markers of cardiovascular risk. Liraglutide is an injectable glucagon-like peptide-1 (GLP-1) analogue which is indicated for treatment of type 2 diabetes in adults. It has been shown to induce weight loss and reduction in insulin resistance in type 2 diabetic and obese patients. Treatment with clinically relevant doses of liraglutide for at least 20 weeks leads to weight loss in obese patients with or without type 2 diabetes. However, there is little information on the effects of GLP-1 analogues on NASH, particularly in comparison to other modalities of weight loss such as surgery.

Our study will also compare the accuracy of magnetic resonance imaging (MRI), the current noninvasive reference standard method for measuring hepatic fat content, with liver biopsy for staging of NASH. Biopsy is the current gold standard, but carries higher procedural risks, and is less convenient and acceptable to patients than non-invasive methods of evaluating severity and activity of NASH. Hence liver biopsy for week 0, 26 and week 52 is optional based on patient consent. We will also measure biomarkers for altered hepatic lipid partitioning and adipokine action, increased oxidative stress and free fatty acid lipotoxicity, which have been implicated in the pathogenesis of NAFLD, and which may be useful non-invasive methods for evaluating the severity of NASH and the efficacy of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 27.5 kg/m2
* Waist circumference (WC) > 90 cm (male) or > 80 cm (female)
* Diagnosis of NASH based on Liver Function Test Results ,Ultrasound Hepato-Biliary System (HBS) findings and / or Liver Biopsy
* HbA1c < 8%* *Subjects in the bariatric surgery arm will not need to fulfil this criterion.

Exclusion Criteria:

* Currently using insulin-sensitising agents (metformin, pioglitazone), weight loss medication (orlistat, phentermine). Patients taking any of these drugs will require a three month washout period before enrolment.
* Pregnancy
* Significant cardiovascular or respiratory disease
* Renal impairment with eGFR < 60 ml/min
* Hepatitis B or C carrier, liver disease other than NAFLD
* History of pancreatitis
* Personal or family history of multiple endocrine neoplasia type 2 or thyroid carcinoma
* Untreated hypothyroidism or hyperthyroidism
* Current psychiatric illness
* Cardiac pacemaker, metallic prosthetic heart valves and other contraindications to MRI scan
* Current smoker
* Alcohol intake ≥ 14 units/week

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in NASH | 12 months
  Reduction/normalization in transaminases, liver fat

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Khoo J, Hsiang JC, Taneja R, Koo SH, Soon GH, Kam CJ, Law NM, Ang TL. Randomized trial comparing effects of weight loss by liraglutide with lifestyle modification in non-alcoholic fatty liver disease. Liver Int. 2019 May;39(5):941-949. doi: 10.1111/liv.14065. Epub 2019 Feb 24. PMID 30721572